CLINICAL TRIAL: NCT03369899
Title: Effectiveness and Safety Study of the FreeStyle Libre Flash Glucose Monitoring System in Pediatric Populations
Brief Title: FreeStyle Libre Flash Glucose Monitoring System in Pediatric Populations
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-17167
Record Dates: First submitted 2017-12-04; First posted 2017-12-12 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-01

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring System — Subjects will wear the FreeStyle Libre Flash Glucose Monitoring System and will receive no treatment except for safety purposes.

SUMMARY:
This study is a non-randomized, single-arm, multi-center study that is designed to evaluate the safety and effectiveness of the FreeStyle Libre Flash Glucose Monitoring Systems in pediatric populations.

DETAILED DESCRIPTION:
Up to 100 subjects will be enrolled at up to six (6) clinical research sites in the United States. Subjects will wear two Sensors. Each Sensor will have a paired Reader that will be given to the subject. All Readers will be masked during the study (i.e. subjects will not be able to view glucose results obtained from the Sensor on the Reader screen). Subjects will be asked to perform at least 4 capillary Blood Glucose (BG) tests per day using the primary Reader. Interstitial glucose readings from each Sensor will be obtained with the corresponding Readers immediately following each BG test. Subjects will be instructed to report any problems with the device. Subjects will make two (2) to five (5) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Based on the subjects age and weight, subjects will have up to two (2) in-clinic visits during which intravenous blood draws and Yellow Springs Instrument (YSI) reference testing will occur.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 4 years of age.
* Subject must have a diagnosis of type 1 or type 2 diabetes mellitus
* Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily).
* Subject must be currently performing at least four (4) capillary blood glucose tests per day.
* Subject is willing to perform a minimum of 4 finger sticks per day during the study.
* If 6 year of age or older and weighing at least 19 kg (41.8 lbs.), willing to allow medical personnel to insert at IV catheter in the arm to allow for venous blood samples to be obtained per the study protocol
* Subject and/or guardian must be able to read and understand English.
* In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* Subject must be available to participate in all study visits.
* Subject must be willing and able to provide written signed and dated informed assent (subjects aged 13 to 17 only).
* Subject's parent, guardian or legally authorized representative must be willing and able to provide written informed consent.

Exclusion Criteria:

* Subject is 18 years of age or older.
* Subject is 6 years or older and weighs less than 19 kg (subjects unable to complete 4 hours of YSI testing).
* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is known to be pregnant or becomes pregnant during the study (applicable to female subjects only).
* Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
* Subject is currently participating in another clinical trial.
* Subject has had significant blood loss within 112 days (3.7 months) prior to the beginning of the study activities subjects.
* Subject is anemic (only applicable to subjects age 6 or older and weighing at least 19 kg) defined as hemoglobin levels below 11.5 g/dL for subjects aged 6-11 years old, less than 12.0 g/dL for subjects aged 12-15 years old, less than 12.0 g/dL for females aged 15-17 and less than 13.0 g/dL for males aged 15-171, or as determined by investigator.
* Subject has X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
* Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects aged 4-17 years, with type 1 or type 2 diabetes who currently perform capillary blood glucose (BG) testing at least four (4) times a day.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
System Performance | Up to 14 days
  System performance will be characterized with respect to YSI reference venous plasma sample measurements for subjects aged 6 and older. Capillary blood glucose (BG) reference will be used for subjects aged less than 6 years of age.
  For subjects age 6 years and older, point accuracy of the system will be evaluated as the proportion of System readings that are within ±20% of the YSI reference value for YSI glucose levels ≥ 80 mg/dL and within ±20 mg/dL for YSI glucose levels <80 mg/dL. For subjects of age less than 6 years, ages 4 and older the system will be evaluated as the proportion of System readings that are within ±20% of the BG reference value for BG glucose levels ≥ 80 mg/dL and within ±20 mg/dL for BG glucose levels <80 mg/dL.
System Related adverse device effects | up to 45 days
  System will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, Ph.D., Study Director — Abbott Diabetes Care
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No